CLINICAL TRIAL: NCT00916812
Title: Hyomental Distance Ratio as a Predictor for Difficult Intubation in Elective and Emergency Cesarean Section.
Brief Title: Sensitivity of Hyomental Distance Ratio as a Single Predictor of Difficult Intubation in Obstetrics
Acronym: HMDR
Status: Completed | Type: Observational
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Collaborators: Corniche Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ACH 0901
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Caesarean Section
Keywords: Difficult intubation; Hyomental distance; Obstetric; Mallampati classification; Thyromental distance; Sternomental distance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a study to detect the sensitivity of thyromental distance ratio as a single predictor for difficult intubation in patients undergoing cesarean section under general anesthesia.

DETAILED DESCRIPTION:
The authors intend to use the HMDR for detection of difficult intubation in parturient undergoing cesarean section that is either elective or emergency.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for cesarean section under general anesthesia

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients presenting for cesarean section under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Prediction of difficult intubation | One year

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad, MD, AB, SB, Principal Investigator — King Khaled Eye Specialist Hospital
Locations (1):
- Al Corniche Hospital, Abu Dhabi, United Arab Emirates